CLINICAL TRIAL: NCT02264574
Title: A Randomized, Multi-center, Open-label, Phase 3 Study of the Bruton's Tyrosine Kinase Inhibitor Ibrutinib in Combination With Obinutuzumab Versus Chlorambucil in Combination With Obinutuzumab in Subjects With Treatment-naïve Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: A Multi-Center Study of Ibrutinib in Combination With Obinutuzumab Versus Chlorambucil in Combination With Obinutuzumab in Patients With Treatment naïve Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1130-CA
Record Dates: First submitted 2014-10-01; First posted 2014-10-15 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small-Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; obinutuzumab; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- IBR + OB (Experimental): Ibrutinib (IBR) given orally at a dose of 420 mg/day until progressive disease or unacceptable toxicity. Intravenous obinutuzumab (OB) given on Days 1 and 2 (100 mg on Day 1 and 900 mg on Day 2), 1000 mg on Days 8 and 15 of Cycle 1 and 1000 mg on Day 1 of each cycle up to 6 cycles or until progressive disease or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Obinutuzumab
- CLB + OB (Experimental): Chlorambucil (CLB) given orally at a dose of 0.5 mg/kg body weight up to a total of 6 cycles on Days 1 and 15 of each cycle or until disease progression or unacceptable toxicity.
  Intravenous obinutuzumab given on Days 1 and 2 (100 mg on Day 1 and 900 mg on Day 2), 1000 mg on Days 8 and 15 of Cycle 1 and 1000 mg on Day 1 of each cycle up to 6 cycles or until disease progression or unacceptable toxicity.
  Interventions: Drug: Obinutuzumab; Drug: Chlorambucil

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be supplied as 140 mg hard gelatin capsules for oral (PO) administration.
  Arms: IBR + OB
Drug: Obinutuzumab — Obinutuzumab will be supplied as 1000 mg/40 mL solution in a single-use vial for intravenous (IV) administration
Drug: Chlorambucil — Chlorambucil will be supplied as 2 mg film-coated tablets for oral (PO) administration
  Arms: CLB + OB

SUMMARY:
The primary objective of this study is to evaluate the efficacy of ibrutinib in combination with obinutuzumab compared to chlorambucil in combination with obinutuzumab based on the Independent Review Committee (IRC) assessment of progression free survival (PFS). Efficacy will be evaluated according to 2008 International Workshop for Chronic Lymphocytic Leukemia (IWCLL) criteria with the modification for treatment-related lymphocytosis, in subjects with treatment-naive CLL or SLL.

ELIGIBILITY:
Inclusion Criteria:

Disease Related:

1. Diagnosis of CLL/SLL that meets IWCLL diagnostic criteria.
2. Age 65 yrs and older OR if less than 65 years, must have at least one of the following criteria:

   * Cumulative Illness Rating Score (CIRS) >6
   * Creatinine clearance estimated <70 mL/min using Cockcroft-Gault equation.
   * Del 17p by fluorescence in situ hybridization (FISH) or TP53 mutation by polymerase chain reaction (PCR) or Next Generation Sequencing
3. Active disease meeting at least 1 of the following IWCLL criteria for requiring treatment:

   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and thrombocytopenia
   * Massive, progressive, or symptomatic splenomegaly
   * Massive nodes (at least 10 cm longest diameter), or progressive or symptomatic lymphadenopathy.
   * Progressive lymphocytosis with an increase of more than 50 percent over a 2-month period or a lymphocyte doubling time (LDT) of <6 months. LDT may be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In patients with initial blood lymphocyte counts of <30,000/µL, LDT should not be used as a single parameter to define indication for treatment. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (eg, infections) should be excluded.
   * Autoimmune hemolytic anemia and/or immune thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy.
   * Autoimmune hemolytic anemia is defined by at least one marker of hemolysis (indirect bilirubin above the upper limit of normal (ULN) not due to liver disease, increased lactate dehydrogenase (above ULN) without alternative etiology, or increased absolute reticulocytosis (above ULN) or bone marrow erythropoiesis in the absence of bleeding AND at least one marker direct or indirect autoimmune mechanism (positive direct antiglobulin for immunoglobulin G [IgG] or C3d, cold agglutinins).
   * Immune thrombocytopenia is defined by platelets ≤100,000/µL and increased megakaryocytes on the bone marrow exam.
   * Constitutional symptoms, defined as one or more of the following disease-related symptoms or signs, documented in the patient's record prior to randomization:
   * unintentional weight loss >10 percent within 6 months prior to screening.
   * significant fatigue (inability to work or perform usual activities).
   * fevers >100.5°F or 38.0°C for 2 or more weeks prior to screening without evidence of infection.
   * night sweats for more than 1 month prior to screening without evidence of infection.
4. Measurable nodal disease by computed tomography (CT), defined as at least 1 lymph node >1.5 cm in the longest diameter in a site that has not been previously irradiated. An irradiated lesion may be assessed for measurable disease only if there has been documented progression in that lesion since radiotherapy has ended.

   Laboratory
5. Adequate hematologic function independent of transfusion and growth factor support for at least 7 days prior to screening and randomization.
6. Adequate hepatic and renal function
7. Men and women ≥ 18 years of age.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Exclusion Criteria:

1. Any prior treatment of CLL or SLL
2. Evidence of central nervous system (CNS) involvement with primary disease of CLL/SLL
3. History of other malignancies, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
4. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura
5. Known or suspected history of Richter's transformation.
6. Concurrent administration of >20mg/day of prednisone within 7 days of randomization unless indicated for prophylaxis or management of allergic reactions (eg, contrast)
7. Known hypersensitivity to one or more study drugs
8. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
9. Any uncontrolled active systemic infection or an infection requiring systemic treatment that was completed ≤ 7 days before randomization.
10. Known bleeding disorders or hemophilia.
11. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
12. Known history of human immunodeficiency virus (HIV) or active with hepatitis B virus (HBV) or hepatitis C virus (HCV).
13. Major surgery within 4 weeks of randomization.
14. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
15. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
16. Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
17. Concomitant use of warfarin or other vitamin K antagonists.
18. Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor.
19. Lactating or pregnant
20. Unwilling or unable to participate in all required study evaluations and procedures.
21. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Styles, Study Director — Pharmacyclics LLC.
Locations (71):
- United States (8):
  - Site Reference ID/Investigator# 0241, La Jolla, California
  - Site Reference ID/Investigator# 0844, Fort Myers, Florida
  - Site Reference ID/Investigator# 0763, West Palm Beach, Florida
  - Site Reference ID/Investigator# 071, Louisville, Kentucky
  - Site Reference ID/Investigator# 0712, Las Vegas, Nevada
  - Site Reference ID/Investigator# 0845, Cincinnati, Ohio
  - Site Reference ID/Investigator# 0868, Chattanooga, Tennessee
  - Site Reference ID/Investigator# 0123, Nashville, Tennessee
- Australia (6):
  - Site Reference ID/Investigator #0503, Woolloongabba, Queensland
  - Site Reference ID/Investigator# 0650, Adelaide, South Australia
  - Site Reference ID/Investigator# 0888, Ballarat, Victoria
  - Site Reference ID/Investigator# 0193, Box Hill, Victoria
  - Site Reference ID/Investigator# 0633, Fitzroy, Victoria
  - Site Reference ID/Investigator# 0170, Heidelberg, Victoria
- Austria (2):
  - Site Reference ID/Investigator# 0352, Linz
  - Site Reference ID/Investigator# 0869, Salzburg
- Belgium (2):
  - Site Reference ID/Investigator# 0559, Leuven
  - Site Reference ID/Investigator# 0850, Turnhout
- Site Reference ID/Investigator# 018, Edmonton, Alberta, Canada
- Czechia (2):
  - Site Reference ID/Investigator# 0564, Hradec Králové
  - Site Reference ID/Investigator# 0854, Prague
- France (4):
  - Site Reference ID/Investigator# 0769, Pessac, Gironde
  - Site Reference ID/Investigator# 0520, Nantes, Loire Atlantique
  - Site Reference ID/Investigator# 0775, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Site Reference ID/Investigator# 0855, Bayonne, Pyrenees Atlantiques
- Israel (6):
  - Site Reference ID/Investigator# 0573, Haifa
  - Site Reference ID/Investigator# 0577, Jerusalem
  - Site Reference ID/Investigator# 0579, Jerusalem
  - Site Reference ID/Investigator# 0575, Petah Tikva
  - Site Reference ID/Investigator# 0856, Tel Aviv
  - Site Reference ID/Investigator# 0875, Ẕerifin
- Italy (8):
  - Site Reference ID/Investigator# 0860, Florence
  - Site Reference ID/Investigator# 0523, Milan
  - Site Reference ID/Investigator# 0581, Milan
  - Site Reference ID/Investigator# 0584, Milan
  - Site Reference ID/Investigator# 0524, Modena
  - Site Reference ID/Investigator# 0582, Novara
  - Site Reference ID/Investigator# 0732, Roma
  - Site Reference ID/Investigator# 0859, Siena
- New Zealand (3):
  - Site Reference ID/Investigator# 0663, Auckland
  - Site Reference ID/Investigator# 662, Auckland
  - Site Reference ID/Investigator# 0586, Hamilton
- Poland (2):
  - Site Reference ID/Investigator# 0592, Brzozów
  - Site Reference ID/Investigator# 0531, Lodz
- Russia (5):
  - Site Reference ID/Investigator# 0708, Nizhny Novgorod
  - Site Reference ID/Investigator# 0707, Ryazan
  - Site Reference ID/Investigator# 0881, Saint Petersburg
  - Site Reference ID/Investigator# 710, Saint Petersburg
  - Site Reference ID/Investigator# 304, Yaroslavl
- Spain (9):
  - Site Reference ID/Investigator# 0604, L'Hospitalet de Llobregat, Madrid
  - Site Reference ID/Investigator# 0536, Majadahonda, Madrid
  - Site Reference ID/Investigator# 0533, Barcelona
  - Site Reference ID/Investigator# 0534, Barcelona
  - Site Reference ID/Investigator# 0535, Barcelona
  - Site Reference ID/Investigator# 0537, Madrid
  - Site Reference ID/Investigator# 0864, Madrid
  - Site Reference ID/Investigator# 0874, Madrid
  - Site Reference ID/Investigator# 0790, Salamanca
- Sweden (4):
  - Site Reference ID/Investigator# 0870, Borås
  - Site Reference ID/Investigator# 0865, Luleå
  - Site Reference ID/Investigator# 0631, Lund
  - Site Reference ID/Investigator# 0632, Stockholm
- Turkey (Türkiye) (6):
  - Site Reference ID/Investigator# 0678, Istanbul, Nisantasi
  - Site Reference ID/Investigator# 0608, Ankara
  - Site Reference ID/Investigator# 606, Ankara
  - Site Reference ID/Investigator# 0889, Denizli
  - Site Reference ID/Investigator# 0601, Izmir
  - Site Reference ID/Investigator# 0866, Samsun
- United Kingdom (3):
  - Site Reference ID/Investigator# 0867, Harlow, Essex
  - Site Reference ID/Investigator# 0365, London
  - Site Reference ID/Investigator# 0543, London

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to individual participant data from clinical studies conducted by Pharmacyclics LLC, an AbbVie Company, can be submitted through Yale Open Data Access (YODA) Project site at the following link.
URL: http://yoda.yale.edu

REFERENCES:
- [Result] Moreno C, Greil R, Demirkan F, Tedeschi A, Anz B, Larratt L, Simkovic M, Samoilova O, Novak J, Ben-Yehuda D, Strugov V, Gill D, Gribben JG, Hsu E, Lih CJ, Zhou C, Clow F, James DF, Styles L, Flinn IW. Ibrutinib plus obinutuzumab versus chlorambucil plus obinutuzumab in first-line treatment of chronic lymphocytic leukaemia (iLLUMINATE): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Jan;20(1):43-56. doi: 10.1016/S1470-2045(18)30788-5. Epub 2018 Dec 3. PMID 30522969
- [Derived] Abuhelwa AY, Almansour SA, Brown JR, Al-Shamsi HO, Abuhelwa Z, Kharaba Z, Bustanji Y, Semreen MH, Ali S, Alhuraiji A, McKinnon RA, Sorich MJ, Alzoubi KH, Hopkins AM. Statin use and survival in CLL/SLL treated with ibrutinib: pooled analysis of 4 randomized controlled trials. Blood Adv. 2025 Jul 22;9(14):3566-3575. doi: 10.1182/bloodadvances.2024015287. PMID 40266025
- [Derived] Moreno C, Greil R, Demirkan F, Tedeschi A, Anz B, Larratt L, Simkovic M, Novak J, Strugov V, Gill D, Gribben JG, Kwei K, Dai S, Hsu E, Dean JP, Flinn IW. First-line treatment of chronic lymphocytic leukemia with ibrutinib plus obinutuzumab versus chlorambucil plus obinutuzumab: final analysis of the randomized, phase III iLLUMINATE trial. Haematologica. 2022 Sep 1;107(9):2108-2120. doi: 10.3324/haematol.2021.279012. PMID 35021599
- [Derived] Burger JA, Robak T, Demirkan F, Bairey O, Moreno C, Simpson D, Munir T, Stevens DA, Dai S, Cheung LWK, Kwei K, Lal I, Hsu E, Kipps TJ, Tedeschi A. Up to 6.5 years (median 4 years) of follow-up of first-line ibrutinib in patients with chronic lymphocytic leukemia/small lymphocytic lymphoma and high-risk genomic features: integrated analysis of two phase 3 studies. Leuk Lymphoma. 2022 Jun;63(6):1375-1386. doi: 10.1080/10428194.2021.2020779. Epub 2022 Jan 11. PMID 35014928
- [Derived] Allan JN, Shanafelt T, Wiestner A, Moreno C, O'Brien SM, Li J, Krigsfeld G, Dean JP, Ahn IE. Long-term efficacy of first-line ibrutinib treatment for chronic lymphocytic leukaemia in patients with TP53 aberrations: a pooled analysis from four clinical trials. Br J Haematol. 2022 Feb;196(4):947-953. doi: 10.1111/bjh.17984. Epub 2021 Dec 5. PMID 34865212
- [Derived] Greil R, Tedeschi A, Moreno C, Anz B, Larratt L, Simkovic M, Gill D, Gribben JG, Flinn IW, Wang Z, Cheung LWK, Nguyen AN, Zhou C, Styles L, Demirkan F. Pretreatment with ibrutinib reduces cytokine secretion and limits the risk of obinutuzumab-induced infusion-related reactions in patients with CLL: analysis from the iLLUMINATE study. Ann Hematol. 2021 Jul;100(7):1733-1742. doi: 10.1007/s00277-021-04536-6. Epub 2021 May 20. PMID 34018029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 71 sites: 8 in the US, 36 in the EU, and 27 sites in 6 additional countries (Canada, Australia, New Zealand, Russia, Israel, Turkey). The first participant consented 06 October 2014. The last visit of the last participant was 03 September 2019, with a final database lock of 17 October 2019.
Pre-assignment Details: Eligible participants were required to have had a diagnosis of active CLL/SLL conformant to IWCLL 2008 criteria. All subjects were required to have measurable nodal disease. Key exclusion criteria included any previous CLL/SLL treatment; known lymphoma or leukemia of the central nervous system, history/current evidence of Richter's transformation.
Groups:
- IBR+OB: Ibrutinib (IBR) given orally at a dose of 420 mg/day until progressive disease or unacceptable toxicity.
  Intravenous obinutuzumab (OB) given on Days 1 and 2 (100 mg on Day 1 and 900 mg on Day 2), 1000 mg on Days 8 and 15 of Cycle 1 and 1000 mg on Day 1 of each cycle up to 6 cycles or until progressive disease or unacceptable toxicity.
- CLB+OB: Chlorambucil (CLB) given orally at a dose of 0.5 mg/kg body weight up to a total of 6 cycles on Days 1 and 15 of each cycle or until disease progression or unacceptable toxicity.
  Intravenous obinutuzumab (OB) given on Days 1 and 2 (100 mg on Day 1 and 900 mg on Day 2), 1000 mg on Days 8 and 15 of Cycle 1 and 1000 mg on Day 1 of each cycle up to 6 cycles or until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | IBR+OB | CLB+OB
Started | 113 | 116
Completed (On-study until study termination by sponsor.) | 84 | 86
Not Completed | 29 | 30
Not completed — Death | 21 | 21
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Other, Not Specified | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IBR+OB | CLB+OB | Total
Number analyzed (Participants) | 113 | 116 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 46
  >=65 years | 91 | 92 | 183
Age, Continuous [Median (Full Range); unit: years] | 70.0 [47 to 87] | 72.0 [40 to 86] | 71.0 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 37 | 83
  Male | 67 | 79 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 109 | 110 | 219
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 2 | 4
  White | 109 | 111 | 220
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
  Czechia | 8 | 6 | 14
  United Kingdom | 2 | 2 | 4
  Spain | 17 | 9 | 26
  Russia | 11 | 9 | 20
  New Zealand | 0 | 9 | 9
  Canada | 3 | 5 | 8
  Austria | 5 | 6 | 11
  Sweden | 8 | 3 | 11
  Turkey | 15 | 13 | 28
  Belgium | 2 | 2 | 4
  Poland | 2 | 2 | 4
  Italy | 13 | 15 | 28
  Israel | 5 | 11 | 16
  France | 3 | 5 | 8
  Australia | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis: Progression Free Survival (PFS) Based on Independent Review Committee (IRC) Assessment - Kaplan Meier Landmark Estimates at Month 30
Description: PFS was defined as time from the date randomization to the date of first IRC-confirmed disease progression (PD) or date of death due to any cause, whichever occurred first, regardless of the use of subsequent antineoplastic therapy prior to documented PD or death. Assessment of PD was conducted in accordance with the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria (Halleck et al) with the modification that treatment-related lymphocytosis in the absence of other signs or symptoms of disease progression was not considered progressive disease.
  The primary analysis was performed after observing 94 PFS events as pre-specified in the study protocol. As the median PFS was not reached in the experimental (IBR+OB) arm at the time of the analysis, Kaplan Meier landmark estimates of the PFS rate at 30 months (that is, the estimated percentage of participants with progression-free survival at Month 30) are presented.
Time Frame: Month 30 (Median follow-up time was 31.3 months at the time of the primary analysis [data cutoff date: 26 March 2018]).
Population: Intent to Treat population: all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 78.5 [69.5 to 85.2] | 31.1 [22.5 to 40.0]
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; To preserve the study wise type I error rate of 0.05, the primary and secondary endpoints were tested based on serial gatekeeping testing procedure at the two-sided significance level of 0.05 according to the hierarchical order of the primary analysis outcome measures presented in this record; Test type: Superiority; p < 0.0001, Log Rank; The treatment effect was tested with an unstratified log rank test; Hazard Ratio (HR) = 0.231, 95% CI 2-sided [0.145 to 0.367] — The hazard ratio and its 95% confidence interval were estimated using a Cox regression model with treatment as the only covariate

2. Secondary Outcome: Primary Analysis: PFS in High-Risk Sub-Population (del17p/TP53 Mutation/Del 11q) Based on IRC Assessment - Kaplan Meier Landmark Estimates at Month 30
Description: PFS was analyzed within the high-risk sub-population of participants with del17p or TP53 mutation or del 11q at baseline per central lab results. PFS was defined as time from the date randomization to the date of first IRC-confirmed PD or date of death due to any cause, whichever occurred first, regardless of the use of subsequent antineoplastic therapy prior to documented PD or death. Assessment of PD was conducted in accordance with the IWCLL 2008 criteria (Halleck et al) with the modification that treatment-related lymphocytosis in the absence of other signs or symptoms of PD was not considered progressive disease.
  As the median PFS was not reached in the experimental (IBR+OB) arm at the time of the analysis, Kaplan Meier landmark estimates of the PFS rate at 30 months (that is, the estimated percentage of participants with progression-free survival at Month 30) are presented.
Time Frame: Month 30 (Median follow-up time was 31.3 months at the time of the primary analysis [data cutoff date: 26 March 2018]).
Population: High-Risk Sub-Population Analysis Set: participants with del17p or TP53 mutation or del 11q at baseline per central lab results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 30 | 45
percentage of participants | 82.4 [62.7 to 92.3] | 14.1 [5.3 to 26.9]
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank; The treatment effect was tested with an unstratified log rank test; Hazard Ratio (HR) = 0.119, 95% CI 2-sided [0.046 to 0.307] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Primary Analysis: Rate of Sustained Hemoglobin Improvement
Description: Percentage of participants with sustained hemoglobin improvement, defined as hemoglobin increase ≥ 2 g/dL over baseline continuously for ≥ 56 days without blood transfusions or growth factors.
Time Frame: Median follow-up time was 31.3 months at the time of the primary analysis (data cutoff date: 26 March 2018).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 39.8 | 44.0
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5253, Chi-squared

4. Secondary Outcome: Primary Analysis: Rate of Minimal Residual Disease (MRD)-Negative Response
Description: Percentage of participants who achieved MRD-negative response, defined as < 1 CLL cell per 10,000 leukocytes as assessed by flow cytometry of a bone marrow aspirate per central laboratory. MRD samples were collected before initiation of subsequent antineoplastic treatment and MRD status was reported by central lab within 5 days after collection date. Participants with missing MRD data were considered non-responders.
Time Frame: Median follow-up time was 31.3 months at the time of the primary analysis (data cutoff date: 26 March 2018).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 20.4 | 17.2
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5465, Chi-squared

5. Secondary Outcome: Primary Analysis: Overall Response Rate (ORR) Based on IRC Assessment
Description: ORR, defined as the percentage of participants achieving a best overall response of protocol-specified complete response (CR), CR with incomplete blood count recovery (CRi), nodular partial response (nPR), or partial response (PR) per IRC assessment at or prior to initiation of subsequent antineoplastic therapy. Assessment of response included physical examination, radiographic imaging, and evaluation of blood and marrow (if applicable), evaluated in accordance with the IWCLL 2008 criteria (Halleck et al). CR, CRi, nPR, and PR required confirmation with 2 consecutive assessments that were at least 56 days apart and no use of blood supportive product and/or growth factor during this period. Kaplan-Meier estimate.
Time Frame: Median follow-up time was 31.3 months at the time of the primary analysis (data cutoff date: 26 March 2018).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 88.5 | 73.3
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0035, Chi-squared; Rate Ratio = 1.208, 95% CI 2-sided [1.062 to 1.373]

6. Secondary Outcome: Primary Analysis: Overall Survival (OS) - Kaplan Meier Landmark Estimates at Month 30
Description: OS, defined as the time from the date of randomization to the date of death from any cause. All deaths observed as the time of the analysis were considered as events. For participants who were not known to have died at the time of the analysis, OS data were censored at the date last known alive.
  As the median OS was not reached in either treatment arm at the time of the analysis, Kaplan Meier landmark estimates of the OS rate (that is, the estimated percentage of participants still surviving at Month 30 [primary analysis]) are presented.
Time Frame: Month 30 (Median follow-up time was 31.3 months at the time of the primary analysis [data cutoff date: 26 March 2018]).
Population: Intent to Treat population: all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 85.5 [77.4 to 90.9] | 84.9 [76.8 to 90.4]
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8057, Log Rank; The treatment effect was tested with an unstratified log rank test; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.479 to 1.772] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Primary Analysis: Rate of Grade ≥ 3 or Serious Infusion-Related Reaction (IRR) Adverse Events
Description: Percentage of participants experiencing grade ≥ 3 (severe or life threatening) or serious IRR adverse events that started on the day of an obinutuzumab infusion and were assessed as related or possibly related to obinutuzumab. Categories included those events with the Medical Dictionary for Regulatory Activities (MedDRA) dictionary preferred term of IRR and those events which are among the customized standardized MedDRA query (SMQ) for IRR.
Time Frame: Median follow-up time was 31.3 months at the time of the primary analysis (data cutoff date: 26 March 2018).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants
  IRR (Preferred Term) | 2.7 | 8.6
  By Customized SMQ | 4.4 | 9.5
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; IRR Preferred Term To preserve the study wise type I error rate of 0.05, the primary and secondary endpoints were tested based on serial gatekeeping testing procedure at the two-sided significance level of 0.05 according to the hierarchical order of the primary analysis outcome measures presented in this record; Test type: Superiority; p = 0.0835, Fisher Exact
Statistical Analysis 2: Comparison: IBR+OB vs CLB+OB; IRR By Customized SMQ To preserve the study wise type I error rate of 0.05, the primary and secondary endpoints were tested based on serial gatekeeping testing procedure at the two-sided significance level of 0.05 according to the hierarchical order of the primary analysis outcome measures presented in this record; Test type: Superiority; p = 0.1944, Fisher Exact

8. Secondary Outcome: Primary Analysis: Rate of Sustained Platelet Improvement
Description: Percentage of participants with platelet counts increase ≥ 50% over baseline continuously for ≥ 56 days without blood transfusion or growth factors.
Time Frame: Median follow-up time was 31.3 months at the time of the primary analysis (data cutoff date: 26 March 2018).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 29.2 | 13.8
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0045, Chi-squared

9. Secondary Outcome: Primary Analysis: Rate of Clinically Meaningful Improvement in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EuroQol Five-Dimension (EQ-5D-5L)
Description: Percentage of participants with EQ-5D-5L utility score increase ≥ 0.08 points over baseline at or prior to initiation of subsequent antineoplastic therapy. The EQ-5D-5L is a standardized non-disease specific instrument for describing and valuing health-related quality of life, comprising 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe the participant's current health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. A unique EQ-5D-5L health state is defined by combining the numeric level scores for each of the 5 dimensions and the total score is normalized from -0.594 to 1.000, with higher scores representing a better health state. An increase in the EQ-5D-5L total score indicates improvement. Participants with missing EQ-5D-5L data were considered not achieving clinically meaningful improvement.
Time Frame: Median follow-up time was 31.3 months at the time of the primary analysis (data cutoff date: 26 March 2018).
Population: Intent to Treat population: all randomized participants with a baseline and post-baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 109 | 107
percentage of participants | 54.9 | 56.0
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8590, Chi-squared

10. Secondary Outcome: Final Analysis: PFS in High-Risk Population (del17p/TP53 Mutation/Del 11q/Unmutated Immunoglobulin Heavy Chain Variable Region [IGHV]) Based on Investigator Assessment - Kaplan Meier Landmark Estimates at Month 48
Description: PFS was analyzed within the high-risk population of participants with del17p or TP53 mutation or del 11q or IGHV unmutated at baseline per central lab results. PFS was defined as time from the date randomization to the date of first investigator-confirmed PD or date of death due to any cause, whichever occurred first, regardless of the use of subsequent antineoplastic therapy prior to documented PD or death. Assessment of PD was conducted in accordance with the IWCLL 2008 criteria (Halleck et al) with the modification that treatment-related lymphocytosis in the absence of other signs or symptoms of PD was not considered progressive disease.
  As the median PFS was not reached in the experimental (IBR+OB) arm at the time of the analysis, Kaplan Meier landmark estimates of the PFS rate at 48 months (that is, the estimated percentage of participants with progression-free survival at Month 48) are presented.
Time Frame: Month 48 (Median follow-up time was 44.6 months at the time of the final analysis [data cutoff date: 17 October 2019]).
Population: High-Risk Population Analysis Set: participants with del17p or TP53 mutation or del 11q or IGHV unmutated at baseline per central lab results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 73 | 75
percentage of participants | 70.3 [57.6 to 79.8] | 8.0 [2.3 to 18.6]
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; Test type: Superiority; p < 0.0001, Log Rank; The treatment effect was tested with an unstratified log rank test; Hazard Ratio (HR) = 0.169, 95% CI 2-sided [0.102 to 0.282] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Final Analysis: Rate of Sustained Hemoglobin Improvement
Description: as for outcome 3
Time Frame: Median follow-up time was 44.6 months at the time of the final analysis (data cutoff date: 17 October 2019).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 44.2 | 44.0
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; Test type: Superiority; p = 0.9657, Chi-squared

12. Secondary Outcome: Final Analysis: Rate of Minimal Residual Disease (MRD)-Negative Response
Description: as for outcome 4
Time Frame: Median follow-up time was 44.6 months at the time of the final analysis (data cutoff date: 17 October 2019).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 24.8 | 17.2
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; Test type: Superiority; p = 0.1612, Chi-squared

13. Secondary Outcome: Final Analysis: ORR Based on Investigator Assessment
Description: ORR, defined as the percentage of participants achieving a best overall response of protocol-specified CR, CRi, nPR or PR per investigator assessment at or prior to initiation of subsequent antineoplastic therapy. Assessment of response included physical examination, radiographic imaging, and evaluation of blood and marrow (if applicable), evaluated in accordance with the IWCLL 2008 criteria (Halleck et al). CR, CRi, nPR, and PR required confirmation with 2 consecutive assessments that were at least 56 days apart and no use of blood supportive product and/or growth factor during this period. Kaplan-Meier estimate.
Time Frame: Median follow-up time was 44.6 months at the time of the final analysis (data cutoff date: 17 October 2019).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 91.2 | 81.0
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; Test type: Superiority; p = 0.0273, Chi-squared; Rate Ratio = 1.125, 95% CI 2-sided [1.013 to 1.250]

14. Secondary Outcome: Final Analysis: Overall Survival (OS) - Kaplan Meier Landmark Estimates at Month 48
Description: OS, defined as the time from the date of randomization to the date of death from any cause. All deaths observed as the time of the analysis were considered as events. For participants who were not known to have died at the time of the analysis, OS data were censored at the date last known alive.
  As the median OS was not reached in either treatment arm at the time of the analysis, Kaplan Meier point estimates of the OS rate (that is, the estimated percentage of participants still surviving at Month 48 [final analysis]) are presented.
Time Frame: Month 48 (Median follow-up time was 44.6 months at the time of the final analysis [data cutoff date: 17 October 2019]).
Population: Intent to Treat population: all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 80.5 [71.6 to 86.9] | 81.3 [72.8 to 87.4]
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; Test type: Superiority; p = 0.7934, Log Rank; The treatment effect was tested with an unstratified log rank test; Hazard Ratio (HR) = 1.083, 95% CI 2-sided [0.595 to 1.973] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Final Analysis: Rate of Sustained Platelet Improvement
Description: as for outcome 8
Time Frame: Median follow-up time was 44.6 months at the time of the final analysis (data cutoff date: 17 October 2019).
Population: Intent to Treat population: all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 30.1 | 14.7
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; Test type: Superiority; p = 0.0050, Chi-squared

16. Primary Outcome: Final Analysis: PFS Based on Investigator Assessment - Kaplan Meier Landmark Estimates at Month 48
Description: PFS was defined as time from the date randomization to the date of first investigator-confirmed PD or date of death due to any cause, whichever occurred first, regardless of the use of subsequent antineoplastic therapy prior to documented PD or death. Assessment of PD was conducted in accordance with the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria (Halleck et al) with the modification that treatment-related lymphocytosis in the absence of other signs or symptoms of disease progression was not considered progressive disease.
  As the median PFS was not reached in the experimental (IBR+OB) arm at the time of the analysis, Kaplan Meier landmark estimates of the PFS rate at 48 months (that is, the estimated percentage of participants with progression-free survival at Month 48) are presented.
Time Frame: Month 48 (Median follow-up time was 44.6 months at the time of the final analysis [data cutoff date: 17 October 2019]).
Population: Intent to Treat population: all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IBR+OB | CLB+OB
Number analyzed (Participants) | 113 | 116
percentage of participants | 74.0 [64.3 to 81.4] | 22.0 [11.0 to 35.4]
Statistical Analysis 1: Comparison: IBR+OB vs CLB+OB; Test type: Superiority; p < 0.0001, Log Rank; The treatment effect was tested with an unstratified log rank test; Hazard Ratio (HR) = 0.251, 95% CI 2-sided [0.162 to 0.389] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug. Median treatment duration for the IBR+OB arm was 42.3 (IBR) and 4.6 (OB) months. Median treatment duration for the CLB+OB arm was 5.1 (CLB) and 4.6 (OB) months. Final analysis data (data cutoff date: 17 October 2019).
Description: One participant in the CLB+OB arm was randomized but went off study without any treatment. This participant had received baseline assessments and was included in all efficacy analyses but was excluded from safety population, i.e. not at risk for adverse event assessment.
Arm/Group | IBR+OB | CLB+OB
All-Cause Mortality (participants affected / at risk) | 22/113 | 21/115
Serious Adverse Events (participants affected / at risk) | 69/113 | 41/115
Other Adverse Events (participants affected / at risk) | 112/113 | 111/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IBR+OB (N=113) | CLB+OB (N=115)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 7
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Catheter site haematoma (General disorders) | 1 | 0
Death (General disorders) | 2 | 0
Multi-organ disorder (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 4
Sudden Death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Infective aneurysm (Infections and infestations) | 1 | 0
Listeria sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 5
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Urosepsis (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 8
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Complete Suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IBR+OB (N=113) | CLB+OB (N=115)
Anaemia (Blood and lymphatic system disorders) | 19 | 29
Increased tendency to bruise (Blood and lymphatic system disorders) | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 50 | 73
Spontaneous haematoma (Blood and lymphatic system disorders) | 10 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 39 | 29
Atrial fibrillation (Cardiac disorders) | 16 | 0
Palpitations (Cardiac disorders) | 7 | 3
Cataract (Eye disorders) | 11 | 1
Dry eye (Eye disorders) | 7 | 3
Lacrimation increased (Eye disorders) | 8 | 5
Vision blurred (Eye disorders) | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Constipation (Gastrointestinal disorders) | 19 | 14
Diarrhea (Gastrointestinal disorders) | 39 | 12
Dyspepsia (Gastrointestinal disorders) | 9 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 15 | 34
Stomatitis (Gastrointestinal disorders) | 7 | 1
Vomiting (Gastrointestinal disorders) | 12 | 14
Asthenia (General disorders) | 12 | 17
Chills (General disorders) | 7 | 10
Fatigue (General disorders) | 22 | 19
Oedema peripheral (General disorders) | 14 | 8
Peripheral swelling (General disorders) | 7 | 2
Pyrexia (General disorders) | 19 | 28
Bronchitis (Infections and infestations) | 8 | 2
Cellulitis (Infections and infestations) | 6 | 3
Conjunctivitis (Infections and infestations) | 12 | 2
Herpes zoster (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 15 | 4
Oral herpes (Infections and infestations) | 1 | 6
Pneumonia (Infections and infestations) | 12 | 5
Respiratory tract infection (Infections and infestations) | 8 | 1
Upper respiratory tract infection (Infections and infestations) | 18 | 7
Urinary tract infection (Infections and infestations) | 13 | 7
Contusion (Injury, poisoning and procedural complications) | 6 | 1
Fall (Injury, poisoning and procedural complications) | 10 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 26 | 61
Blood creatine increased (Investigations) | 8 | 1
Weight decreased (Investigations) | 3 | 6
Decreased appetite (Metabolism and nutrition disorders) | 11 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 15 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2
Iron deficiency (Metabolism and nutrition disorders) | 9 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 10
Dizziness (Nervous system disorders) | 12 | 7
Headache (Nervous system disorders) | 9 | 13
Tremor (Nervous system disorders) | 4 | 7
Anxiety (Psychiatric disorders) | 10 | 8
Depression (Psychiatric disorders) | 7 | 1
Insomnia (Psychiatric disorders) | 13 | 5
Haematuria (Renal and urinary disorders) | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 7 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 7 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 4
Rash (Skin and subcutaneous tissue disorders) | 10 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 2
Hypertension (Vascular disorders) | 22 | 5
Hypotension (Vascular disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until the earlier of (i) results of study are submitted for publication (ii) notification that submission of the multicenter results are no longer planned (iii) 18 months after study termination.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT02264574/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT02264574/SAP_001.pdf